CLINICAL TRIAL: NCT07154862
Title: Membrane Sweeping as an Induction Method and Maternal Experience: a Phenomenological Qualitative Study
Acronym: Sweep
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Preziosi Jessica, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7350
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-02

CONDITIONS: Membrane Stripping; Patient Experience; Labour, Induced; Phenomenology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This qualitative phenomenological study explores women's experiences with membrane sweeping, a common mechanical method of labor induction. Membrane sweeping is considered a low-cost and low-risk procedure recommended by several guidelines, including NICE, before proceeding to pharmacological or mechanical induction. Despite its widespread use, little evidence is available regarding how women perceive and experience this procedure.

In this single-center, prospective observational study, women with low-risk singleton pregnancies between 40+0 and 41+2 weeks of gestation will be recruited at the "Oltretermine" outpatient clinic of Fondazione Policlinico Universitario Agostino Gemelli, Rome. After providing informed consent, participants who undergo membrane sweeping will be invited to take part in a semi-structured interview within 48-72 hours postpartum during hospital stay.

The primary objective is to describe women's lived experiences of membrane sweeping at term. Secondary objectives include describing women's sociodemographic and obstetric characteristics and their overall birth experience. Data will be analyzed thematically to identify recurring concepts and themes.

This study is independent, non-funded, and will enroll approximately 12-20 women, until data saturation is reached. All procedures comply with the Declaration of Helsinki, GDPR, and national privacy regulations.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >18 and ≤40 years
* Women with singleton pregnancy
* Women with cephalic presentation
* Women able to read and understand the Italian language
* Women with gestational age between 40+0 and 41+2 weeks
* Signed informed consent provided by the participant

Exclusion Criteria:

* Women younger than 18 years or older than 40 years
* Women unable to read and understand the Italian language

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nulliparous and multiparous women aged 18-40 years, with singleton cephalic pregnancies at 40+0 to 41+2 weeks of gestation, receiving care at the "Oltretermine" outpatient clinic of Fondazione Policlinico Universitario Agostino Gemelli, Rome. Participants must be able to read and understand Italian and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Lived experience of membrane sweeping | Within 48-72 hours after childbirth
  Qualitative description of women's perceptions, feelings, and overall experience related to membrane sweeping at term. Data will be collected through semi-structured interviews and analyzed thematically.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Direction, Roma, Italy